CLINICAL TRIAL: NCT04982731
Title: Developing and Evaluating a Positive Assurance Intervention on Recovery Outcomes in mTBI Patients
Brief Title: Positive Assurance and mTBI
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: University of Arkansas, Fayetteville (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: U20-05-4050
Record Dates: First submitted 2021-04-07; First posted 2021-07-29 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: MTBI - Mild Traumatic Brain Injury; Concussion, Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Assurance Discharge Video Educational Intervention (EDUC). (Experimental): The video intervention will be administered to participants that are randomly assigned to the EDUC group. In addition, current standard of care discharge instructions will also be provided to the participant. This EDUC intervention will consist of a brief, three to five-minute informative video message from the clinical neuropsychologist at the Inova Sports Medicine Concussion Program. Participants will be instructed to view the video at least once every 24 - 48 hours prior to their visit to the concussion clinic.
  Interventions: Other: Positive Assurance
- Standard of Care Instructions (Treatment as Usual: TAU ) (No Intervention): The Acute Concussion Evaluation (ACE) Care plan in place at the Inova PED/GoHealth Urgent Care sites is the standard-of-care discharge instruction for individuals with mTBI. This care plan provides patient and caregiver education about mTBI and emphasizes the monitoring of symptoms, signs of deterioration that may warrant urgent medical attention, and encourages the patient to follow up with their physician for follow up. Participants who are randomized into the TAU group will receive this standard of care treatment in video format, however these participants will not be given a QR code to watch the intervention video.

INTERVENTIONS:
Other: Positive Assurance — Positive assurance is a low-cost, non-pharmacological strategy commonly used by specialty clinics to manage anxiety in individuals with mTBI. Positive assurance is comprised of words of affirmation given to individuals with a medical condition by a healthcare provider that are centered on hope and positive recovery expectations (i.e., "You will recover," "This can be treated").
  Arms: Positive Assurance Discharge Video Educational Intervention (EDUC).

SUMMARY:
This study will develop and validate a new educational video that provides positive assurance about mild traumatic brain injury (mTBI) recovery for patients with mTBI.

DETAILED DESCRIPTION:
The research team will investigate the effect of this new Positive Assurance discharge intervention video on state anxiety and clinical recovery outcomes in patients with mTBI. A sample of adolescent and young adult patients (13-21yrs) will be recruited for participation that present with a potential mTBI diagnosis and receive specialty referral to the Inova Sports Medicine Concussion Program for follow-up care. Investigators will employ a randomized controlled trial (RCT) to enroll two groups of mTBI patients: 1) a group that receives the video intervention (EDUC), and 2) a group that receives standard discharge instructions (i.e., treatment as usual: TAU).

ELIGIBILITY:
COHORT 1 (no longer being recruited):

INCLUSION CRITERIA:

Subjects must meet the following criteria in order to be eligible to participate:

1. 13-21 years
2. Has sustained an external force to head or body resulting in neurological symptoms and at least one reported symptom is attributed to the mTBI (e.g., dizziness, confusion, headache, postural instability, light/noise sensitivity, nausea)
3. Has receive a medical diagnosis of mTBI from an emergency physical at the IFH Pediatrics ED or Inova-GoHealth Urgent Care clinic within 72 hours of injury
4. Is able to provide remote informed written consent (parent) and assent

EXCLUSION CRITERIA:

Subjects who meet any of the following criteria will not be eligible to participate:

1. Loss of consciousness > 30 minutes in conjunction with the injury
2. Glasgow Coma Scale (GCS) score < 13
3. Has sustained a previous mTBI within the past 6 months
4. Has a neurological disorder (e.g., epilepsy)
5. Has a positive finding on brain imaging (e.g., CT, MRI) that suggests a severe closed head or open injury involving any structural damage or abnormality (e.g., fracture, subdural hematoma)
6. Has a previous history of neurosurgery
7. Does not speak English as a primary language
8. Requires admission to the hospital
9. Has developmental delays
10. Prisoner
11. Pregnant*
12. Has been previously enrolled in the study
13. Members of same household will not be included as they may determine their group assignment if more than one person from same household is included and assigned to different groups.

COHORT 2:

INCLUSION CRITERIA:

Subjects must meet the following criteria in order to be eligible to participate:

1. 13-21 years
2. Has scheduled an appointment to be evaluated at the Inova Sports Medicine Concussion Clinic for a traumatic closed head injury that has occurred within the past 30 days
3. The time between study enrollment and the initial clinical visit is at least two days
4. Is able to provide remote informed written consent (parent) and assent

EXCLUSION CRITERIA:

Subjects who meet any of the following criteria will not be eligible to participate:

1. Loss of consciousness > 30 minutes in conjunction with the injury
2. Glasgow Coma Scale (GCS) score < 13
3. Has sustained a previous mTBI within the past 6 months
4. Has a neurological disorder (e.g., epilepsy)
5. Has a positive finding on brain imaging (e.g., CT, MRI) that suggests a severe closed head or open injury involving any structural damage or abnormality (e.g., fracture, subdural hematoma)
6. Has a previous history of neurosurgery
7. Does not speak English as a primary language
8. Requires admission to the hospital
9. Has developmental delays
10. Prisoner
11. Pregnant*
12. Has been previously enrolled in the study
13. Members of same household will not be included as they may determine their group assignment if more than one person from same household is included and assigned to different groups.

WITHDRAWAL CRITERIA (BOTH COHORTS):

1. Upon examination, if the clinical team determines that a participant did not sustain/cannot confirm a concussion, the subject will be withdrawn from the study.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 229 (Estimated)
Dates: Start 2021-10-15 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Behavioral Regulation Assessment for Concussion (BRAC) | Gathered at Baseline Visit
  The Behavioral Regulation Assessment for Concussion (BRAC) is a five-item, four-point Likert scale (with values ranging from '0-Never' to '5-Most of the Time') assessment for the frequency of self-reported behavioral regulation behaviors that occurred during the past seven days. Scores range from 0 to 20, with higher scores indicating a better outcome. Likert scale scores are reported for each item, with a higher score indicating greater frequency. An average score for the BRAC is the average of all the scores across the items.
Expectations of Recovery Scale | Gathered at Baseline Visit
  The Expectations of Recovery Scale will be used to measure the effect of positive assurance on recovery. This is a seven-item scale that asks individuals to assess whether they think they will get better soon, return to usual activities/work within the next month, return to the pre-injury performance and to consider what they had been told about their injury and what those closest to them advised. Items within this scale are scored independently of each other, therefore neither higher nor lower scores indicate a better or worse outcome.

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | Gathered at Baseline Visit and through study completion, an average of one month
  The State-Trait Anxiety Inventory (STAI) will be used to assess state anxiety in participants ages 15 years and older. The S-Anxiety scale (STAI Form Y-1) consists of twenty statements that are rated on a four-point Likert scale (1- not at all; 4 - very much so) that evaluate how respondents feel "right now, at this moment." The T-Anxiety scale (STAI Form Y-2) consists of twenty statements rated on a four-point Likert scale (1- almost never; 4 - almost always) that assess how people generally feel. Scores for both scales are continuous and range from 20-80, and clinical levels of state anxiety are classified with scores >40.
mTBI Symptoms | Gathered at Baseline Visit and through study completion, an average of one month
  The Post-Concussion Symptom Scale (PCSS) will be used to assess mTBI symptoms. This measure includes 22 symptoms (e.g., headache, nausea, dizziness, etc…) that are rated by the patient on a seven-point Likert scale (e.g., 0 = mild, 6 = severe). Outcome scores for the PCSS are total number of reported symptoms (0 - 22) and total symptom severity score (0 - 132).
Immediate Post-concussion Assessment and Cognitive Test (ImPACT) | Gathered at Baseline Visit and through study completion, an average of one month
  Investigators will assess cognitive function using the Immediate Post-concussion Assessment and Cognitive Test (ImPACT) computerized tool. ImPACT assesses attention, visual working memory, verbal recognition memory, reaction time, visual processing speed, numerical sequencing ability, and learning.
Vestibular/Ocular Motor Screening (VOMS) | Gathered at Baseline Visit and through study completion
  Investigators will use the Vestibular/Ocular Motor Screening (VOMS) tool to assess vestibular and ocular motor impairment via patient-reported symptom provocation. The VOMS consists of the following five components: 1) smooth pursuits, 2) horizontal and vertical saccades, 3) convergence, 4) horizontal and vertical vestibular ocular reflex (VOR) and 5) visual motion sensitivity (VMS). Self-reported symptom severities (0-10) are reported with each of the five components, with higher ratings reflecting greater symptom severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Inova Health System, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: No